CLINICAL TRIAL: NCT05956730
Title: Audio-guided Home Physical Activity to Support People With Low Vision: Physical Performance and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2422
Record Dates: First submitted 2023-03-23; First posted 2023-07-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Low Vision Blindness
Keywords: Physical Activity; Physical Performance; Quality of Life
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The proposed protocol includes a part of aerobic training and a subsequent part of strengthening exercises for large muscle groups. The total duration of each session will be approximately 30 minutes. There are 2 weekly training sessions for 3 months.
  Interventions: Other: Physical Activity (AUD)
- Group 2 (Active Comparator): The proposed protocol includes a part of aerobic training and a subsequent part of strengthening exercises for large muscle groups. The total duration of each session will be approximately 30 minutes. There are 2 weekly training sessions for 3 months.
  Interventions: Other: Physical Activity (SUP)

INTERVENTIONS:
Other: Physical Activity (AUD) — Home training of patients with severe low vision managed through audio-guides (AUD).
  Arms: Group 1
Other: Physical Activity (SUP) — Training of patients with severe low vision in a gym supervised by a personal trainer (SUP).
  Arms: Group 2

SUMMARY:
The aim of the project is to investigate the effectiveness of a home training managed through audio-guides in comparison to a classic supervised training on the physical and psychological parameters of patients with severe low vision.

In this study the feasibility and effectiveness of a self-managed physical activity protocol with audio guides on physical performance (strength, mobility and aerobic capacity) will be assessed and compared to the same protocol supervised in a fitness environment.

Secondary aims are the effects of the two types of administration of the protocol on quality of life, autonomy and psychological impact on the caregiver.

DETAILED DESCRIPTION:
According to the World Health Organization, low vision is that condition of permanent reduction of the visual function which does not allow an individual to fully develop his relationship activity, conduct a normal work activity, pursue his needs and aspirations of life. The increase in life expectancy on the one hand and the increasingly better ability to prevent and treat serious eye diseases, has led in industrialized countries to extraordinarily high numbers of patients who develop serious hypovision in adulthood or advanced age.

Since regular physical activity is essential for maintaining good health in older adults, even those with limited mobility, to maintain muscle mass and good balance (thus preventing falls) the use of audio devices or workouts carried out through audio guides for management of exercises in autonomy and at home will be tested. The aim of the project is to investigate the effectiveness of a home training protocol managed through audio-guides, in comparison to a classic supervised training, on the physical and psychological parameters of patients with severe low vision.

Participants (people with severe low vision) will be randomized into two groups: "audio" group (AUD), trained through exercises explained through audio files and "supervised" group (SUP), trained in a gym supervised by a personal trainer.

The training protocol will have a total duration of 3 months, with 2 weekly sessions and a monthly re-planning of loads and intensities.

The participants of the SUP group will be trained at the Adapted Motor Activity Laboratory (LAMA) of the University of Pavia.

To evaluate the changes induced by exercise, subjects will undergo physical tests and questionnaires, at the beginning and monthly until the end of the study.

It is expected that combined training should increase aerobic capacity and general strength of the individual, as well as have a positive effect on quality of life and psychosocial life, both using audio-guided and supervised training.

Obtaining these benefits with a self-managed training strategy would lead to greater independence of the subject and would expand the possibility of intervention in the population with low vision. Ultimately, these benefits could also be reflected in the management of the person with low vision by the caregiver and close family members.

ELIGIBILITY:
Inclusion Criteria:

* Residual visus up to 1/10 or residual binocular perimeter less than 30% (Severely visually impaired);
* age greater than or equal to 50 years;
* sedentary lifestyle, PASIPD questionnaire value less than 13.2 Mets hours/day;
* sedentary lifestyle, IPAQ-SF questionnaire value less than 700 Mets/week;
* absence of autonomous mobility with white cane.
* proprioceptive and balance skills such as to allow the protocol to be managed independently and safely, value of the Berg Balance Scale test greater than 35.

Exclusion Criteria:

Subjects who report habitual physical activity or sports;

* PASIPD questionnaire value greater than 13.2 Mets hours/day.
* Subjects at high risk of falling, with a Berg Balance Scale test value of less than 35.
* Subjects with pathologies that are not compatible with carrying out the physical activity protocol in safety and autonomy.-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Timed up and go - version for the visually impaired (TUG-LV) | 3 months
  Assessment of functional walking ability. In this version for patients with visual impairments, the subject must get up from the chair and walk 6 meters to a luminous point (light point) and go back to sit down as quickly as possible.

SECONDARY OUTCOMES:
Sit to stand test (1-MSTS) | 3 months
  Functional evaluation of muscle power. Sitting on a chair without armrests (about 50cm high) and with his hands on his chest, the patient must get up and sit down as quickly as possible, as many times as possible within 1 minute.
Sit and reach test (SR) | 3 months
  Flexibility of the subject's posterior muscle kinetic chain. The subject seated with legs extended on the floor, with bare feet resting on a specific graduated cube, exhales and slowly bends the torso forward (without bending the knees) and tries to reach the farthest point of the cube with his own fingers.
3 minutes step test (3MST) | 3 months
  Assessment of aerobic capacity. Using a 15 cm high step (step), the subject is asked to go up and down the step as many times as possible in 3 minutes. The correct repetitions are recorded, i.e. when in the transition from the ground to the step and vice versa, both feet are on the ground and the knees are extended.
hand-grip test | 3 months
  assessment of generic strength (isometric specification of the hand flexors). The subject seated with his elbow resting on the table (respecting the angles between the bust and forearm according to the guidelines) squeezes a dynamometer with as much force as possible.
Berg Balance Scale | 3 months
  assessment of proprioceptive and balance skills through the execution of dynamic movements and the maintenance of static postures, in order to obtain information on the subject's motor skills, on the possible need for walking aids and on the risk of fall it presents
Satisfaction Profile (SAT-P) questionnaire | 3 months
  level of personal satisfaction and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Pavia, Italy

REFERENCES:
- [Derived] Correale L, Schmid M, Decortes F, Martinis L, Liberali G, Bandirali L, Cusella G, Montomoli C. Audio-guided exercise at home: Preliminary findings from a pilot study on physical activity for people with low vision. PM R. 2026 Jan 10. doi: 10.1002/pmrj.70081. Online ahead of print. PMID 41518011